CLINICAL TRIAL: NCT03252990
Title: Molecular Imaging of Coronary Plaque Vulnerability Using 18F-fluorocholine PET-MRI in Patients With Coronary Artery Disease
Brief Title: 18F-fluorocholine PET-MR Imaging of Coronary Plaque Vulnerability
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: VieCuri Medical Centre (Other); Stichting de Weijerhorst (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL58752.068.16
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Myocardial Infarction; Myocardial Ischemia; Atherosclerosis; Coronary Artery Disease; Coronary Stenosis; Heart Attack; Multi Vessel Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Atherosclerosis; Coronary Artery Disease; Coronary Stenosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Optimization subjects: Before the enrollment of the actual study subjects, 5 stable angina pectoris patients that are scheduled for a PCI procedure at the MUMC+ will be included at the MUMC+ for a single PET-MRI scan to optimize the parameters of the coronary PET-MRI scan. All patients will receive standard, guideline-based clinical care, while PET-MRI will be performed as an additional measurement.
  Interventions: Diagnostic Test: PET-MRI
- Patients from the VieCuri hospital: 15 NSTEMI or STEMI patients who underwent urgent percutaneous coronary intervention (PCI) of the culprit vessel, who are diagnosed with multivessel coronary disease and are currently scheduled for a second PCI at the VieCuri hospital will be included. These patients will be subjected to an additional 18F-choline PET-MRI examination at the MUMC+ and an additional optical coherence tomography (OCT) examination (during the PCI procedure) at the Viecuri hospital. OCT will be performed as a reference standard to validate 18F-choline PET-MRI for detection of vulnerable plaques in the coronary arteries. All patients will receive standard, guideline-based clinical care, while PET-MRI and OCT will be performed as additional measurements.
  Interventions: Diagnostic Test: PET-MRI; Procedure: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: PET-MRI — Additional 18F-choline PET-MRI examination
Procedure: Optical Coherence Tomography — Additional optical coherence tomography (OCT) examination (during the already planned routine PCI procedure)
  Groups: Patients from the VieCuri hospital

SUMMARY:
This study is designed as a prospective observational feasibility study. The investigators will study whether vulnerable plaques on OCT (fibrous cap ≤ 70 μm) show a locally increased uptake of 18F-choline on PET-MRI compared to stable plaques and whether the culprit plaque shows a locally increased uptake of 18F-choline on PET-MRI compared to non-culprit plaques. First, 15 NSTEMI or STEMI patients who underwent urgent percutaneous coronary intervention (PCI) of the culprit vessel, who are diagnosed with multivessel coronary disease and are currently scheduled for a second PCI at the VieCuri hospital will be included. These patients will be subjected to an additional 18F-choline PET-MRI examination at the MUMC+ and an additional optical coherence tomography (OCT) examination (during the PCI procedure at the Viecuri hospital). OCT will be performed as a reference standard to validate 18F-choline PET-MRI for detection of vulnerable plaques in the coronary arteries. In addition, 15 NSTEMI patients, who are scheduled for PCI of the culprit lesion at the MUMC+, will be subjected to an additional 18F-choline PET-MRI examination at the MUMC+. Hereby, the culprit coronary vessel and thereby the culprit plaque can be identified by the location of the myocardial infarct, as identified by late enhanced MRI. The investigators will study whether the culprit plaque shows an increased 18F-choline uptake on 18F-choline PET-MRI compared to non-culprit plaques in the other coronary arteries. All patients will receive standard, guideline-based clinical care, while PET-MRI and OCT will be performed as additional measurements. Before the start of the study, 5 stable angina pectoris patients that are scheduled for a PCI procedure at the MUMC+ will be included at the MUMC+ for a single PET-MRI scan to optimize the parameters of the coronary PET-MRI scan.

DETAILED DESCRIPTION:
Background of the study:

Myocardial infarction (MI) frequently recurs after MI, which may be related to insufficient vulnerable plaque identification using invasive coronary angiography. More accurate identification of vulnerable plaques may improve therapeutic strategies and clinical outcome. Recently, the investigators demonstrated that 18F-choline PET can be used to identify vulnerable carotid plaques. The investigators hypothesize that fully integrated 18F-choline PET-MRI enables detection of vulnerable coronary plaques.

Objective of the study:

The objective is to study the feasibility to detect vulnerable coronary plaques with 18F-choline PET-MRI.

Primary study parameters/outcome of the study:

* To investigate whether vulnerable plaques on OCT (fibrous cap ≤ 70 μm) show a locally increased uptake of 18F-choline on PET-MRI compared to stable plaques.
* To investigate whether the culprit plaque shows a locally increased uptake of 18F-choline on PET-MRI compared to non-culprit plaques.

Secondary study parameters/outcome of the study (if applicable):

* To study whether there is a correlation between the uptake of 18F-choline in coronary plaques and the degree of stenosis as shown on the angiogram acquired during the PCI procedure
* To study whether there is a correlation between the uptake of 18F-choline in coronary plaques and the presence of macrophages, micro-calcifications, lipid-rich necrotic core on OCT
* To investigate whether there is an association between the uptake of 18F-choline in the coronary arteries and that in the carotid arteries.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

This study will not delay any necessary treatment and the study is not expected to adversely affect outcome. The patients from the VieCuri will need to visit the MUMC for the additional PET-MRI scan. All patients in this study, including the 5 patients for protocol optimisation, will receive an average radiation dose of 5.3 mSv (0.019 mSv/MBq [see attachment 1], 280 MBq, average body weight 70 kg) and a maximum radiation dose of 6.8 mSv (360 MBq, ≥ 90 kg body weight) from the 18F-choline tracer. PET-MRI, Gadolinium and 18F-choline are safe and the risk of adverse effects are low (as described in chapter 7). The additional OCT examination is performed during the PCI procedure (only in the 15 patients of the VieCuri hospital), that is part of standard patient care, and carries the same risks as the PCI procedure, including: coronary dissection, air embolism, coronary thrombus, contrast nephropathy, contrast allergy, cardiovascular event, and death (extremely rare). These risks will be minimized by the use of heparin to achieve an Activating Clotting Time (ACT) value of 300, taking care of meticulous positioning of the wire and using the OCT catheter under fluoroscopy guidance. Approximately 15% of the amount of contrast agent that is used during an PCI procedure will be additionally administered during the OCT procedure and 30 seconds of additional fluoroscopy guidance with associated increase in ionizing radiation dose will be used for positioning of the OCT catheter. During the additional PET- MRI and OCT examinations, there is a chance on accidental medical findings. These findings will be reported to the treating physician and the general practitioner of the patient. Study results are expected to contribute to improvement of vulnerable plaque detection for future patients.

ELIGIBILITY:
Group 1 - Protocol optimization: only additional PET-MRI

* Diagnosed with stable angina pectoris and scheduled for a PCI procedure at the MUMC
* Minimum age of 18 years
* Mentally competent
* Having provided informed written consent

Group 2 - Patients included at Viecuri hospital: additional PET-MRI and OCT

* NSTEMI or STEMI patients who underwent urgent percutaneous coronary intervention (PCI) of the culprit vessel, who are diagnosed with multivessel coronary disease and are currently scheduled for a second PCI at the VieCuri hospital
* Currently stable and scheduled for another PCI at the VieCuri hospital to stent another coronary vessel
* Able to visit the MUMC by own transport / train for PET-MR imaging before the new PCI procedure
* Minimum age of 18 years
* Mentally competent
* Having provided informed written consent

Group 3 - Patients included at MUMC+: additional PET-MRI

* Recently diagnosed with NSTEMI and scheduled for a PCI at the MUMC
* GRACE risk score between 90 and 140
* Acute Coronary Syndrome (ACS) type 1
* Minimum age of 18 years
* Mentally competent
* Having provided informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See 'Group descriptions'
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
To investigate whether vulnerable plaques on OCT (fibrous cap ≤ 70 μm) show a locally increased uptake of 18F-choline on PET-MRI compared to stable plaques. | 72 hours
To investigate whether the culprit plaque shows a locally increased uptake of 18F-choline on PET-MRI compared to non-culprit plaques. | 72 hours

SECONDARY OUTCOMES:
To study whether there is a correlation between the uptake of 18F-choline in coronary plaques and the degree of stenosis as shown on the angiogram acquired during the PCI procedure | 72 hours
To study whether there is a correlation between the uptake of 18F-choline in coronary plaques and the presence of macrophages, micro-calcifications, lipid-rich necrotic core on OCT | 72 hours
To investigate whether there is an association between the uptake of 18F-choline in the coronary arteries and that in the carotid arteries. | 1.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No